CLINICAL TRIAL: NCT05548959
Title: Differences in Nycthemeral IOP Variation and Outflow Facility After Filtering Microshunt Versus Canal-Based Ab Interno Glaucoma Surgery
Brief Title: Outflow Facility AIT vs Microshunt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114/21me
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma
Keywords: outflow facility; microshunt; ab interno trabeculectomy; pneumatonometer; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microshunt patients (Experimental): Pneumatonometry of the intraocular pressure was performed on patients who have undergone previous microshunt implantation.
  Interventions: Diagnostic Test: Pneumatonometry after microshunt implantation
- Ab interno trabeculectomy patientes (Experimental): Pneumatonometry of the intraocular pressure was performed on patients who have undergone previous ab interno trabeculectomy.
  Interventions: Diagnostic Test: Pneumatonometry after ab interno trabeculectomy

INTERVENTIONS:
Diagnostic Test: Pneumatonometry after microshunt implantation — Pneumatonometry was perfomed over 24 hours at 5 point in time (5 AM, 11 AM, 4 PM, 8 PM, and midnight) using a Pneumatonometer. The measurement was conducted in the habitual position.
  Arms: Microshunt patients
Diagnostic Test: Pneumatonometry after ab interno trabeculectomy — Pneumatonometry was perfomed over 24 hours at 5 point in time (5 AM, 11 AM, 4 PM, 8 PM, and midnight) using a Pneumatonometer. The measurement was conducted in the habitual position.
  Arms: Ab interno trabeculectomy patientes

SUMMARY:
The purpose of this study was to asses differences in nycthemeral (24-h) intraocular pressure (IOP) profiles and outflow facilities between patients who have undergone epibulbar microshunt implantation and ab interno trabeculectomy, respectively.

DETAILED DESCRIPTION:
Recent studies involving continuous, 24-hour intraocular pressure (IOP) monitoring in glaucoma patients linked IOP variation to disease progression.

No study has previously compared the postoperative IOP variation of microshunt (Preserflo, P) implantation to ab interno trabeculectomy (Trabectome, T).

In this prospective cohort, the investigators analyzed 68 patients (34 P and 34 T) who presented for 24-hour IOP monitoring 6 to 12 months after surgery. Surgery must have been conducted between October 2020 and July 2021. Patients were assigned to each study group according to the intervention undergone, P or T. IOP and tonographic outflow facility were measured in the habitual position using a pneumatonometer. The IOP variation was considered the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have undergone microshunt implantation or ab interno trabeculectomy between 6-12 months ago
* patients suffering from open-angle glaucoma

Exclusion Criteria:

* Patients that have undergone microshunt implantation or ab interno trabeculectomy less than 6 months or over 12 months ago
* patients suffering from angle-closure glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure variation | Obtained 6-12 months after patients have undergone microshunt implantation and ab interno trabeculectomy, respectively. Measurements were taken at 5 points in time over 24 hours (at 5 AM, 11 AM, 4 PM, 8 PM, and midnight).
  24-hour variation in intraocular pressure obtained by the use of a pneumatonometer.

SECONDARY OUTCOMES:
Outflow facility | Obtained 6-12 months after patients have undergone microshunt implantation and ab interno trabeculectomy, respectively. Measurements were taken at 5 points in time over 24 hours (at 5 AM, 11 AM, 4 PM, 8 PM, and midnight).
  Outflow facility of the aqueous humor from the eye obtained by pneumatonography.
Intraocular pressure | Obtained 6-12 months after patients have undergone microshunt implantation and ab interno trabeculectomy, respectively. Measurements were taken at 5 points in time over 24 hours (at 5 AM, 11 AM, 4 PM, 8 PM, and midnight).
  Intraocular pressure obtained by the use of a Pneumatonometer

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology University Hospital Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Deployed Pneumatonometer Device — https://www.reichert.com/en/products/model-30